CLINICAL TRIAL: NCT00890851
Title: Evaluation of Procedure Tuna Within the Framework of a Hospitalization of Short Duration
Brief Title: Procedure Transurethral Needle Ablation (TUNA) and Hospitalization of Short Duration
Acronym: EPURE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Mathieu Quintin, Department of clinical research and development
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P050302
Record Dates: First submitted 2009-04-29; First posted 2009-04-30 (Estimated); Last update posted 2009-10-01 (Estimated); Status verified 2009-04

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: Radiofrequency; Mini invasin surgery; Outpatient treatment; Men health
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Transurethral Resection of Prostate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Procedure TUNA (Other)
  Interventions: Procedure: Transurethral Needle Ablation (TUNA)

INTERVENTIONS:
Procedure: Transurethral Needle Ablation (TUNA) — Transurethral needle ablation of benign prostatic hyperplasia by radio frequencies
  Other Names: radiofrenquency prostate

SUMMARY:
The TUNA is a known and already old technique. There exists, in the literature, a certain number of studies showing the long-term effectiveness (5 years), evaluated on the IPS and the flow mictional.This effectiveness is slightly lower than that of the endoscopic resection of prostate. This technique does not present the disadvantages of the surgery prostate sufferer on ejaculation. Moreover, it can be carried out in short hospitalization or ambulatory as it is the case in particular in the States Unis. The aim of the study which will be led by the AP-HP will be thus to test the feasibility of the TUNA during a hospitalization of less 24 hours.

DETAILED DESCRIPTION:
The TUNA is a known and already old technique. There exists, in the literature, a certain number of studies showing the long-term effectiveness (5 years), evaluated on the IPS and the flow mictional. This effectiveness is slightly lower than that of the endoscopic resection of prostate. This technique does not present the disadvantages of the surgery prostate sufferer on ejaculation. Moreover, it can be carried out in short hospitalization or ambulatory as it is the case in particular in the States Unis. The aim of the study which will be led by the AP-HP will be thus to test the feasibility of the TUNA during a hospitalization of less the 24h.

Objective one: To test the feasibility of a procedure TUNA at the time of a hospitalization of less 24h.

Number of patients: A sample of N=70 patients will make it possible to estimate the frequency of success with a precision of ± 10% for any frequency higher than 75%.

Analyse statistical: Principal analyze: Count held of the aim of the study the principal analyses will be descriptives. For the variables qualitative or semi-quantitative bilateral the confidence frequencies and their interval at 95% (IC95) will be presented. If the conditions of use of the asymptotic estimators would not be filled, of the exact estimators will be used. For the quantitative averages and IC95%, median variables and outdistances interquartile will be calculated. Together analyses will be presented for the general population and by center.

Secondary analyze: In case of rate of important failure, an exploratory analysis at end of identification of the predictive factors of failure will be made by analysis in multivariate logistic regression.

Awaited results: The precise evaluation carried out by the present study will make it possible to evaluate the benefit report/ratio risks in the short run procedure and its feasibility within the framework of a hospitalization in surgery ambulatory. The implications are important. Indeed, if this technique can be done into ambulatory with a high rate of success, then this technique of treatment could be proposed in alternative of the medical treatment or to the bad responders with the medical treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Man whose age is superior or egal to 45 and inferior or egal to 85 years
2. Patient presenting an anaesthetic risk of ASA 1 at 3
3. Patient accepting the protocol, in particular the return to residence with a sounder
4. Patient presenting a TUBA related to a HBP and lasting since more than 3 months

   1. with a gene score higher superior or egal to 3
   2. with a score IPS superior to 8
5. Patient presenting a prostate whose estimated weight is inferior or egal to 80g, without median lobe prevailing and whose transverse width lies between 34 and 80 mm.
6. Patient having a residue post mictional lower than 200cc.
7. Patient presenting a normal renal function
8. Patient having a result PSA £ 4 ng/ml, or negative biopsies if PSA > 4 and < 10 ng/ml
9. Patient having given his free and in writing lit assent
10. Patient affiliated to the Social security or an assimilated mode
11. Patient having stopped his treatment by 5 alpha reductase since at least a month (1)

Exclusion Criteria:

1. Patient presenting a urinary infection
2. Patient presenting an acute retention of urine
3. Patient presenting a neurological bladder and/or of an anomaly of the sphincter
4. Patient currently under anticoagulant treatment.
5. Patient currently under anti-inflammatory treatment.
6. Patient presenting an affection or a confirmed or suspected malignant tumour of the prostates or vegie.
7. Patient presenting an antecedent of surgery prostatic
8. Patient presenting of the biopsies prostate sufferers carried out less than 4 months before procedure TUNA
9. Patient introducing of the antecedents of vesical lithiasis, haematuria important, contracting of the urethra, stenosis of the vesical collar, pathologies of the bladder or sweetened diabetes affecting vesical operation,
10. Patient presenting a prosthesis in the zone being able to be affected by the procedure
11. Patient presenting a desire of fertility
12. Patient presenting an anorectal pathology
13. Patient presenting an allergy to the anaesthesia locale
14. Patient whose follow-up seems incompatible with the needs for the study

Ages: 45 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2006-03; Primary Completion 2008-12 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Left the hospital | the evening of the intervention
Not hospitalized for a complication related to the intervention | in the month following the intervention

SECONDARY OUTCOMES:
Evaluation of the satisfaction of the intervention for the patient | at 1 month
Evaluation for the micturition of the following parameters | at 1 month
Evaluation of the appeared minor complications | at 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand LUKACS, MD,PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital TENON - Service d'Urologie, Paris, France